CLINICAL TRIAL: NCT02999360
Title: Aerobic Exercise and Aphasia Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-00960
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Aphasia
Keywords: Aphasia; Speech Therapy; Aerobic Exercise (AE)
MeSH Terms: conditions — Aphasia; Communication Disorders | interventions — Language Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment 1 (Experimental)
  Interventions: Behavioral: Language therapy; Behavioral: Background Music; Behavioral: Aerobic Exercise
- Treatment 2 (Active Comparator)
  Interventions: Behavioral: Language therapy; Behavioral: Background Music; Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Language therapy — There will be three blocks of treatment, ideally three times a week 100 minutes per day. Treatment will target impairment-directed speech language therapy (SLT) approaches or compensatory-directed SLT in each of the three treatment blocks. Half of the participants will receive the impairment-directed SLT. Half of the participants, will receive treatment that will target compensatory-directed speech language therapy approaches that are focused on functional communication skills in the conversational context. Methods of treatment will include PACE (Promoting Aphasics Communicative Effectiveness (Davis, 2005), conversational coaching (Hopper et al., 2002), and supported conversation (Kagan et al., 2001). The clinician will model and encourage all (verbal and non verbal) modalities of communication.
Behavioral: Background Music — 30 minutes background music only
Behavioral: Aerobic Exercise — There will be three blocks of treatment and the AE will take place for all participants during one or two treatment blocks (randomly assigned), threetimes a week (sessions are three times a week prior to speech therapy but may be one or two times a week if a session is missed or may be up to four or five times a week if one or two sessions are missed and rescheduled due to weather or other circumstances).
  Other Names: AE

SUMMARY:
The purpose of the study is to determine if speech therapy can be enhanced by Aerobic Exercise (AE). Investigators will use a single subject design to determine if aphasia therapy result in greater gains when combined with aerobic exercise.

DETAILED DESCRIPTION:
Aim 1: To test the feasibility of a research study that combines speech therapy with aerobic exercise (AE). Participants will be alternately assigned to receiving AE during during a 30 minute break from speech therapy.

Aim 2: To test the preliminary efficacy of combining speech therapy with AE to promote language improvements in aphasia. These data will inform the design of a large, controlled clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Aphasia severity based on Western Aphasia Battery-Revised (WAB-R) aphasia quotient(AQ)>50. An AQ of 51-75 correlates to moderate aphasia severity and an AQ of 76 and above correlates to mild aphasia severity. Only participants with mild to moderate aphasia (WAB AQ>50) will be included. The Aphasia Quotient (AQ) is an essential summary value of the individual's aphasic deficit and is proportional to the severity of aphasia regardless of the type of aphasia or etiology of aphasia. Type of aphasia is not an inclusionary/exclusionary criterion because the focus is on language recovery regardless of aphasia type.
* The inclusionary criterion regarding etiology is aphasia post ischemic stroke; no specific location of stroke is required.
* Associated cognitive deficits are not a part of the inclusionary/exclusionary criteria because aphasia is a language disorder and the treatment is a language treatment.
* English is primary language (patient report). Participant may have exposure to another language however English is the native language and primary language used for communication premorbidly.
* At least 9 months post CVA (patient report and confirmed by medical records review when records available). The participant must be at least 9 months post stroke, which is considered to be the chronic stage therefore there is no restriction on the maximum number of months/years post stroke.
* Able to participate in AE based on MD screening that follows recommendations for exercise in stroke patients .
* Have a history of only one stroke.
* Independent in walking (with or without assistive device).
* Medically stable.
* No previous myocardial infarction.
* No significant musculo-skeletal problems from conditions other than stroke.
* History taken by MD and is part of practices standard of care/best practice for physicians interviewing patients.

Exclusion Criteria:

* MD considers participant unable to comply with study requirements.
* MD evaluates medication history and determines if current medications will have a negative impact and if so MD will not recommend patient inclusion.
* Mood will first be screened by the Beck Depression Inventory screen and then assessed with the Beck Depression Inventory (BDI) if the participant does not pass the screening. This is a 21-item self-report assessment designed specifically to identify depression. The items are scored 0 (no problem) to 3. Thus, the possible score is between 0 - 63. A score of 9 or lower is the usual threshold to separate depressed from non-depressed subjects. If a subject scores 10 or higher the subject will not be included in the study and the MD will discuss with the subject the possibility of a referral for a psychiatric evaluation.
* Stroke due to intracranial hemorrhage primarily due to bleeding from ruptured aneurysm or arteriovenous malformation.
* Progressive stroke (primary progressive aphasia diagnosis)
* Comorbid neurological diagnosis (e.g. MS, PD, dementia)
* Unable to perform the required exercises due to a) medical, b) musculo-skeletal, or c) neurological problems (for details see below, a-c)

  1. medical problems: unstable cardiovascular condition, or other serious cardiac conditions (for example, anyone meeting New York Heart Association Class IV criteria, hospitalization for myocardial infarction or heart surgery within 120 days, severe cardiomyopathy or documented serious and unstable cardiac arrhythmias)
  2. musculo-skeletal problems: restricted passive range of motion in the major lower limb joints (that is, an extension deficit of >20° for the affected hip or knee joints, or a dorsiflexion deficit of >20° for the affected ankle)
  3. neurological problems: severity of stroke-related deficits Required help of at least 1 person to walk before stroke due to neurological (for example, advanced Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis) or non-neurological (for example, heart failure, orthopaedic problems) co-morbidities with life expectancy of less than 1 year as determined by physician.
* Drug or alcohol addiction within the last 6 months.
* Significant current psychiatric illness defined as affective disorder unresponsive to medication or bipolar affective disorder, psychosis, schizophrenia or suicidality.
* Current participation in another interventional trial.

Vulnerable Subjects

* People in this study will have mild to moderate aphasia. Although they have language problems aphasia is not an intellectual disorder and patient's aphasia will not be severe. Subjects will have the capacity to consent to participate.

ed deficits Required help of at least 1 person to walk before stroke due to neurological (for example, advanced Parkinson's disease, amyotrophic lateral sclerosis, multiple sclerosis) or non-neurological (for example, heart failure, orthopaedic problems) co-morbidities with life expectancy of less than 1 year as determined by physician.

* Drug or alcohol addiction within the last 6 months.
* Significant current psychiatric illness defined as affective disorder unresponsive to medication or bipolar affective disorder, psychosis, schizophrenia or suicidality.
* Current participation in another interventional trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
The Aphasia Communication Outcome Measure (ACOM) (Hula et al., 2015) | 24 Weeks
  Patient-reported outcome measure of communicative functioning for persons with aphasia
The Boston Naming Test | 24 Weeks
  The examiner begins with Item 1 and continues through Item 60, unless the patient is in distress or refuses to continue. The patient is told to tell the examiner the name of each picture and is given about 20 seconds to respond for each trial. The examiner writes down the patient's responses in detail, using codes. If the patient fails to give the correct response, the examiner at her or his discretion may give the patient a phonemic cue, which is the initial sound of the target word. After the patient completes the test, the examiner scores each item + or - according to the response coding and scoring procedures

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Galletta, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided